CLINICAL TRIAL: NCT06183268
Title: Evaluation of Radiobiological Effects in Skin Toxicities for Head and Neck Cancer Patients With Pencil Beam Scanning Proton Therapy
Brief Title: Evaluation of Radiobiological Effects in Skin Toxicities Head and Neck Cancer Patients With PBS Proton Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Covenant Health Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-484 INV
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Head and Neck Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Radiation: Spot Delete — The treatments plans will utilize the scripted spot delete method to remove spots from the skin rind. To ensure all relevant skin spots are removed, the "SkinSpots" structure will be a 0.5 cm rind extending inward from the skin contour within 5 cm of the CTV. Spots will be removed from this structure and optimization will continue. Optimization objectives will be utilized to spare the skin rind structure during treatment planning, in addition to deleting spots.

SUMMARY:
This purpose of this study is to examine skin reactions (called radiation dermatitis) that occur during pencil beam scanning (PBS) proton therapy. The researchers will test a unique technique called "Spot Delete" to see if it can reduce skin reactions for head & neck patients treated with PBS. The investigators will also use a special computer model to study how the energy of the proton beam (linear energy transfer) is related to these skin reactions. The study involves creating a treatment plan based on a CT scan, which helps guide the proton beam in the body.

DETAILED DESCRIPTION:
This purpose of this study is to examine skin reactions (called radiation dermatitis) that occur during pencil beam scanning (PBS) proton therapy. The researchers will test a unique technique called "Spot Delete" to see if it can reduce skin reactions for head & neck patients treated with PBS. The investigators will also use a special computer model to study how the energy of the proton beam (linear energy transfer) is related to these skin reactions. The study involves creating a treatment plan based on a CT scan, which helps guide the proton beam in the body. The clinical team uses this CT scan to find the best placement for the protons. The "Spot Delete" method prevents protons from stopping in the skin, which is thought to increase skin dose and thus risk and magnitude of radiation dermatitis. During the study, digital photos of patients' skin will be taken to assess the amount of dermatitis (redness, blistering, or peeling). Patients will be given a self-report questionnaire and medical staff will document the skin reactions in the patients' medical charts. The degree of skin reactions will be compared against historical occurrence rates, and the location of any skin reactions that occur will be compared against the predicted location from the computer model. This study carries the same risks as regular proton therapy. Proton therapy, like other cancer treatments, may cause side effects. Some common side effects include skin reactions (such as redness, dryness, itching, blistering, or peeling) in the treatment area. It is important to note that the "Spot Delete" technique aims to specifically address the skin reactions, so there might be a potential reduction in this particular risk.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to be in the study and must have signed an approved consent form conforming to federal and institutional guidelines.
* Patients must be ≥ 18 years old.
* Patient must have biopsy-proven squamous cell carcinoma, originating in the oral cavity, larynx, oropharynx, nasopharynx, or hypopharynx
* Carcinoma of the neck of unknown primary site origin may be included if p16 positive
* Clinical stage T1-2, N0-1, N2a-N3 or T3-4, any N (AJCC, 7th ed.), including no distant metastases
* Patient can have prior surgical resection of a primary cancer in the head and neck at any previous time
* Previous or concurrent chemotherapy is allowed
* No serious health conditions as determined by physician that would impact ability to complete treatment or impact skin in the area of treatment

Exclusion Criteria:

* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Head and neck radiotherapy that does NOT include at least one cervical lymph node level (I, II, III, IV, or V) in the target volume.
* Children
* Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-01-02 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
"Spot Delete: Technique in Proton Therapy Reduces Radiation Dermatitis in Head and Neck Cancer Patients. | Weekly Assessments over 10 weeks, 1 month and 6 months post treatment
  Aim to test the hypothesis that the "Spot Delete" technique in proton therapy reduces radiation dermatitis in head & neck cancer patients compared to historical data from patients who underwent regular proton therapy without the technique. To evaluate this, the investigators will compare the extent of skin reactions in patients who receive proton therapy with the "Spot Delete" technique to historical data from patients who did not receive this treatment.

SECONDARY OUTCOMES:
To investigate how the linear energy transfer (LET) of the proton beam is related to skin reactions. | comparisons to be conducted over a 5 year period
  It is unknown if there is a correlation between the LET lines and the observed skin reactions. To answer this question, LET will be calculated using RayStation for each patient enrolled in the study. The skin reactions' location and severity will be compared with the calculated LET values, allowing researchers to determine any correlation between LET and skin reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Hedrick, PhD, DABR, Principal Investigator — Thompson Proton Center, Director of Medical Physics
Locations (1):
- Thompson Proton Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No